CLINICAL TRIAL: NCT02090634
Title: Texting to Improve Adherence in HIV+ With Bipolar Disorder
Acronym: iTAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, David J. Moore, Ph.D., Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IDEA Award ID09-SD-047
Record Dates: First submitted 2014-03-07; First posted 2014-03-18 (Estimated); Results first posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: HIV Disease; Bipolar Disorder
Keywords: HIV; Bipolar Disorder; Medication Adherence
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Bipolar Disorder; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Personalized Reminder Texting + Psychoeducation (iTAB) (Experimental): Participants in the individualized Texting for Adherence Building (iTAB) arm will receive daily text messaging reminders for antiretroviral and psychotropic medication adherence. These text messages will be targeted to the specific schedule and needs of the individual. Participants will also receive a text message that assesses mood. Finally, participants will receive a one-time psychoeducational intervention reviewing the importance of adherence to anti-HIV and psychotropic medications.
  Interventions: Behavioral: Psychoeducation; Behavioral: individualized Texting for Adherence Building (iTAB)
- Psychoeducation (CTRL) (Active Comparator): Participants will receive a one-time psychoeducational intervention reviewing the importance of adherence to anti-HIV and psychotropic medications. They will also receive daily text messages to assess mood, but these messages will not receive the medication reminder text messages.
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Psychoeducation — Participants will also receive daily text messages to evaluate mood, but these messages will not remind participants about medication adherence.
Behavioral: individualized Texting for Adherence Building (iTAB) — Intervention is designed to send automated text messages to HIV+ persons who have bipolar disorder (BD+). Text messages are personalized, automated, real-time text messages. The iTAB intervention is designed to improve adherence to ART and psychotropic medications among HIV+/BD+ persons above and beyond an active comparator group.
  Arms: Personalized Reminder Texting + Psychoeducation (iTAB)

SUMMARY:
Adherence to combination antiretroviral therapy (ART) is critical for successful HIV viral suppression. Nonadherence to ART poses several potentially serious health consequences, including higher viral loads, faster progression to AIDS, and a heightened risk of viral mutations, treatment resistance and HIV transmission.

The prevalence of serious mental illness (SMI) conditions, including bipolar disorder (BD), is elevated among HIV-infected populations and is associated with poor ART adherence. HIV-infected individuals with co-occurring BD (HIV+/BD+), when compared to demographically similar HIV+/BD- persons, demonstrated poorer ART and psychotropic medication adherence and were twice as likely to be non adherent to their ART regimen using a ≥ 90% cutoff score. HIV+/BD+ individuals are particularly at-risk for medication non adherence, and there is a critical need to develop interventions to improve adherence in this population.

Poor psychotropic medication adherence is also common among people with SMI - it has been estimated that 40% of those with BD do not take their mood stabilizer as prescribed. Among persons with BD, nonadherence to psychotropic medications can lead to greater risk for manic and depressive episodes, decreased quality of life, suicide attempts, and hospitalization.

The utilization of mobile health (i.e., mHealth) technologies to improve everyday functioning is growing. mHealth interventions capitalize on technology already incorporated into most people's daily lives (e.g., cell phones) to assist people with behavior modification and disease self-management. Text messaging, in particular, may support daily ART adherence by delivering reminders at precise times to match an individuals' dosing schedule. The initial evidence for using text messaging to improve ART medication adherence has been compelling. Researchers and clinicians have also started employing technology-based approaches to improve treatment for individuals with BD.

Taken together, a distinct need for RCTs utilizing text messaging to improve medication adherence within an at-risk HIV population is warranted. Individualized Texting for Adherence Building (iTAB) is one such intervention.

The investigators propose an intervention development study designed to address these potential mechanisms of nonadherence with the following Specific Aims: 1) To further develop and refine a personalized, automated, real-time, mobile phone, text messaging intervention (iTAB) designed to improve adherence to ART and psychotropic medications among HIV+/BD+ persons; 2) To evaluate the acceptability and effectiveness of a brief psychoeducation plus text messaging intervention (iTAB) as compared to psychoeducation alone (CTRL) for the improvement of objectively measured medication adherence among HIV+/BD+ persons; and 3) To examine predictors of within-person trajectories of nonadherence using the longitudinal data collected over the study. In order to realize these aims, the investigators will leverage the infrastructure of two unique UCSD resources increasing likelihood of study success, impact, and innovation: 1) the HIV Neurobehavioral Research Program (HNRP), which encompasses multiple NIH-funded studies that focus on the effects of HIV infection, and 2) the California Institute for Telecommunications and Information Technology (Calit2), which conducts research on state-of-the-art wireless means of health promotion. Initially, the investigators will refine the iTAB intervention to ensure that it is user-centered and tailored to the needs of HIV+/BD+ persons via focus groups and rapid prototyping. Once refined, the proposed iTAB intervention will use text messages that are automated, scalable, personalized, interactive, flexible, and motivating. The investigators will assess the acceptability and effectiveness of iTAB in improving objectively measured adherence (i.e., MEMS caps) over a 4-week period via a pilot RCT with 58 participants were randomized into 2 groups (30 HIV+/BD+ assigned to the iTAB intervention and 28 HIV+/BD+ assigned to a psychoeducational control). Predictors of nonadherence including neuropsychological impairment, and mood will be examined to determine whether iTAB is better able to compensate for these factors associated with nonadherence as compared to CTRL. Further refinement to the iTAB intervention will be made in order to pursue a large-scale R01 using the investigators tailored intervention.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* 18 years or older at the time of enrollment
* HIV-infected
* DSM-IV diagnosis Bipolar Disorder
* Taking at least one medication to treat HIV illness
* Taking at least one medication to treat bipolar disorder
* Indication of less than 100% adherence to antiretroviral (ART) medication
* Willingness to use electronic monitoring caps to track ART medication and BD medication
* Willingness to respond to text messages

Exclusion Criteria:

* Axis I psychiatric diagnosis of psychotic spectrum disorder (e.g., schizophrenia)
* Presence of a neurological condition (beyond HIV infection) known to impact cognitive functioning (e.g., Huntington's Disease, Stroke)
* Unwillingness or inability to use electronic medication monitoring technology
* Unwillingness or inability to use daily texting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2010-04; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J Moore, Ph.D., Principal Investigator — University of California, San Diego
Locations (1):
- HIV Neurobehavioral Research Program (HNRP), Department of Psychiatry, Univeristy of California, San Diego, California, United States

REFERENCES:
- [Result] Moore DJ, Poquette A, Casaletto KB, Gouaux B, Montoya JL, Posada C, Rooney AS, Badiee J, Deutsch R, Letendre SL, Depp CA, Grant I, Atkinson JH; HIV Neurobehavioral Research Program (HNRP) Group. Individualized texting for adherence building (iTAB): improving antiretroviral dose timing among HIV-infected persons with co-occurring bipolar disorder. AIDS Behav. 2015 Mar;19(3):459-71. doi: 10.1007/s10461-014-0971-0. PMID 25504449

RESULTS

PARTICIPANT FLOW:
Recruitment Details: HIV+/BD+ participants were recruited from ongoing studies at the UCSD HIV Neurobehavioral Research Program (HNRP).
Pre-assignment Details: 62 participants were assessed for eligibility, and 4 participants were excluded prior to randomization; 2 did not meet study criteria, 2 withdrew. 58 participants were enrolled and randomized into iTAB (n=30) or control group (n=28). 50 participants completed the study and were included in analyses; excluded from analyses were 5 iTAB participants (3 lost MEMS, 2 had adverse events unrelated to study participation) and 3 control participants (1 lost MEMS, 1 lost contact, 1 was deceased).
Groups:
- Personalized Reminder Texting + Psychoeducation (iTAB): Individualized Texting for Adherence Building (iTAB): Participants will receive daily text messaging reminders for antiretroviral and psychotropic medication adherence. These text messages will be targeted to the specific schedule and needs of the individual.
  Psychoeducation: Participants will receive a one-time psychoeducational intervention reviewing the importance of adherence to anti-HIV and psychotropic medications. Participants will also receive daily text messages to assess mood
- Psychoeducation (CTRL): Participants will receive a one-time psychoeducational intervention reviewing the importance of adherence to antiretroviral and psychotropic medications. Participants will also receive daily text messages to assess mood, but these messages will not receive the medication reminder text messages.
Period: Overall Study
Arm/Group | Personalized Reminder Texting + Psychoeducation (iTAB) | Psychoeducation (CTRL)
Started | 30 | 28
Completed | 25 | 25
Not Completed | 5 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Death | 0 | 1
Not completed — Protocol Violation | 3 | 1
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Population: 62 participants were assessed for eligibility; 2 were ineligible and 2 declined to participate. 58 participants were enrolled & randomized to the CTRL (n=28) or iTAB intervention arm (n=30). Analyses included 25 iTAB participants (excluded: 3 lost MEMS, 1 entered rehab facility, 1 had illness & went off meds), and 25 CTRL participants (excluded: 1 lost MEMS, 1 lost contact, 1 deceased unrelated to study).
Groups:
- Personalized Reminder Texting + Psychoeducation (iTAB): The individualized Texting for Adherence Building (iTAB) intervention is designed to improve adherence to antiretroviral and psychotropic medications for HIV+ persons who have bipolar disorder using automated text message reminders. These text messages will be targeted to the specific medication schedule and needs of the individual. Participants will also receive daily text messages to assesses mood. Additionally, participants will receive a one-time psychoeducational intervention reviewing the importance of adherence to antiretroviral and psychotropic medications.
- Psychoeducation (CTRL): HIV+ persons who have bipolar disorder will receive a one-time psychoeducational intervention reviewing the importance of adherence to antiretroviral and psychotropic medications. Participants will also receive daily text messages to assess mood, but these participants will not receive the medication reminder text messages.
- Total: Total of all reporting groups
Arm/Group | Personalized Reminder Texting + Psychoeducation (iTAB) | Psychoeducation (CTRL) | Total
Number analyzed (Participants) | 30 | 28 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 58 participants were enrolled & randomized to the CTRL (n=28) or iTAB intervention arm (n=30). Analyses included 25 iTAB participants (excluded: 3 lost MEMS, 1 entered rehab facility, 1 had illness & went off meds), and 25 CTRL participants (excluded: 1 lost MEMS, 1 lost contact, 1 deceased unrelated to study).
  years
    number analyzed (Participants) | 25 | 25 | 50
    (all) | 48.4 (9.2) | 45.9 (10.2) | 47.1 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 58 participants were enrolled & randomized to the CTRL (n=28) or iTAB intervention arm (n=30). Analyses included 25 iTAB participants (excluded: 3 lost MEMS, 1 entered rehab facility, 1 had illness & went off meds), and 25 CTRL participants (excluded: 1 lost MEMS, 1 lost contact, 1 deceased unrelated to study).
  Participants
    number analyzed (Participants) | 25 | 25 | 50
    Female | 2 | 4 | 6
    Male | 23 | 21 | 44
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: 62 participants were assessed for eligibility; 2 were ineligible and 2 declined to participate. participants were enrolled & randomized to the CTRL (n=28) or iTAB intervention arm (n=30). Analyses included 25 iTAB participants (excluded: 3 lost MEMS, 1 entered rehab facility, 1 had illness & went off meds), and 25 CTRL participants (excluded: 1 lost MEMS, 1 lost contact, 1 deceased unrelated to study).
  Participants
    Non-Hispanic White: number analyzed (Participants) | 25 | 25 | 50
    Non-Hispanic White | 16 | 11 | 27
    Non-Hispanic Black: number analyzed (Participants) | 25 | 25 | 50
    Non-Hispanic Black | 7 | 6 | 13
    Hispanic: number analyzed (Participants) | 25 | 25 | 50
    Hispanic | 2 | 5 | 7
    Hispanic Black: number analyzed (Participants) | 25 | 25 | 50
    Hispanic Black | 0 | 2 | 2
    Native American: number analyzed (Participants) | 25 | 25 | 50
    Native American | 0 | 1 | 1
Region of Enrollment [Number; unit: participants] — Population: Participants were enrolled & randomized to the CTRL (n=28) or iTAB intervention arm (n=30). Analyses included 25 iTAB participants (excluded: 3 lost MEMS, 1 entered rehab facility, 1 had illness & went off meds), and 25 CTRL participants (excluded: 1 lost MEMS, 1 lost contact, 1 deceased unrelated to study).
  participants
    United States: number analyzed (Participants) | 25 | 25 | 50
    United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Proportion Adherent to ARV and Psychotropic Medication by Electronic Monitoring System (MEMS)
Description: MEMS-derived percent adherence to HIV and psychotropic medications over the study period, i.e., ([# of bottle openings]/[# of prescribed doses]*100%).
Time Frame: 4-week
Population: Of the 30 participants in iTAB intervention group, 25 were analyzed; 3 lost MEMS cap, 1 in rehabilitation facility, 1 too sick.Of the 28 participants in CTRL group, 25 were analyzed; 1 lost MEMS cap, 1 lost to follow up, 1 deceased.
Measure: Median (Inter-Quartile Range); unit: percentage of taken doses
Groups:
- Psychoeducation (CTRL): Participants will receive a one-time psychoeducational intervention reviewing the importance of adherence to anti-HIV and psychotropic medications. Participants will also receive daily text messages to assess mood, but these messages will not receive the medication reminder text messages.
Arm/Group | Personalized Reminder Texting + Psychoeducation (iTAB) | Psychoeducation (CTRL)
Number analyzed (Participants) | 25 | 25
percentage of taken doses
  ARV adherence | 90.3 [75.8 to 96.5] | 90.0 [77.6 to 93.3]
  PSY adherence | 83.9 [70.2 to 95.1] | 90.0 [74.5 to 96.7]
Statistical Analysis 1: Comparison: Personalized Reminder Texting + Psychoeducation (iTAB) vs Psychoeducation (CTRL); We conducted Wilcoxon rank sum (Mann-Whitney) tests in order to examine group (i.e., iTAB vs. CTRL) differences on overall adherence to ARV medications; Test type: Superiority; p = 0.95, Wilcoxon (Mann-Whitney) — Cliff's d = 0.01; calculated to estimate the effect size for between-group comparisons with non-parametric data
Statistical Analysis 2: Comparison: Personalized Reminder Texting + Psychoeducation (iTAB) vs Psychoeducation (CTRL); We conducted Wilcoxon rank sum (Mann-Whitney) tests in order to examine group (i.e., iTAB vs. CTRL) differences on overall adherence to PSY medications; Test type: Superiority; p = 0.43, Wilcoxon (Mann-Whitney); Cliff's d = -0.13; calculated to estimate the effect size for between-group comparisons with non-parametric data

2. Primary Outcome: Dose Timing for ARV and Psychotropic Medications as Determined by Electronic Medication Monitoring System (MEMS).
Description: Medication "dose timing window" for participants was calculated by subtracting the time at which the MEMS cap was opened (i.e., dose taken) from the previously indicated targeted time for dosing (i.e., the time at which participants received adherence text messages for the iTAB intervention group, or time at which participants indicated they would take their medication for the control group). Dose timing windows were used in analyses to indicate the discrepancy between intended dosing time and actual dosing time (in minutes) such that higher values indicate more variable dosing (i.e., decreased therapeutic coverage).
Time Frame: 4-week
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: minutes from dosing target time
Arm/Group | Personalized Reminder Texting + Psychoeducation (iTAB) | Psychoeducation (CTRL)
Number analyzed (Participants) | 25 | 25
minutes from dosing target time
  Dose timing window for ART | 27.8 [15.0 to 105.5] | 77.0 [36.3 to 137.8]
  Dose timing window for PST | 46.8 [18.7 to 121.3] | 66.5 [24.0 to 135.0]
Statistical Analysis 1: Comparison: Personalized Reminder Texting + Psychoeducation (iTAB) vs Psychoeducation (CTRL); We conducted Wilcoxon rank sum (Mann-Whitney) tests in order to examine group (i.e., iTAB vs. CTRL) differences on overall dose timing windows for ARV medications; Test type: Superiority; p = 0.02, Wilcoxon (Mann-Whitney) — Cliff's d = 0.37; calculated to estimate the effect size for between-group comparisons with non-parametric data
Statistical Analysis 2: Comparison: Personalized Reminder Texting + Psychoeducation (iTAB) vs Psychoeducation (CTRL); We conducted Wilcoxon rank sum (Mann-Whitney) tests in order to examine group (i.e., iTAB vs. CTRL) differences on overall dose timing windows for PSY medications; Test type: Superiority; p = 0.42, Wilcoxon (Mann-Whitney) — Cliff's d = 0.14; calculated to estimate the effect size for between-group comparisons with non-parametric data

ADVERSE EVENTS:
Arm/Group | Personalized Reminder Texting + Psychoeducation (iTAB) | Psychoeducation (CTRL)
All-Cause Mortality (participants affected / at risk) | 0/30 | 1/28
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/28
Other Adverse Events (participants affected / at risk) | 2/30 | 0/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Personalized Reminder Texting + Psychoeducation (iTAB) (N=30) | Psychoeducation (CTRL) (N=28)
Rehabilitation Facility (Social circumstances) | 1 (1) | 0 (0) — Unrelated to study participation, one participant did not complete the study due to admission to a Rehabilitation Facility
Participant sickness (Immune system disorders) | 1 (1) | 0 (0) — Unrelated to study participation, one participant did not complete the study due to sickness resulting from cessation of medications

LIMITATIONS AND CAVEATS:
1) Small sample size; 2) Short time period; 3) MEMS adherence data based on # of cap openings, not directly whether the medication was ingested; 4) No group without psychoeducation component

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No